CLINICAL TRIAL: NCT05385614
Title: Efficacy of Gamified Cognitive Control Training Using de:)Press on Depression Severity add-on to Treatment as Usual
Acronym: de-press-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 950/2021BO2
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Depression; Cognitive Impairment; Cognitive Dysfunction; Depressive Disorder
MeSH Terms: conditions — Depression; Cognitive Dysfunction; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group that will receive the app after primary endpoint was assessed.
- Intervention (Experimental): Experimental group that will receive the app at the start of their participation
  Interventions: Behavioral: de:)press

INTERVENTIONS:
Behavioral: de:)press — Patients will receive de:)press for the duration of six weeks. They will be encourages to use the app at least three times a week, up to once per day.
  Arms: Intervention

SUMMARY:
Depression is one of the most frequent and devastating psychiatric diseases with a substantial bur-den for patients and society. It is specifically associated with dysfunctional activity in brain networks subserving cognitive control of emotional information processing. Normalization of this activity is a hallmark of various treatment approaches. Computerized training of cognitive control has shown antidepressant effects in experimental lab settings and small clinical pilot trials. However, motiva-tion, treatment adherence, and access for patients are major challenges that limit its broader use. To address these challenges, we developed a software application (de:)press®) that integrates gamification elements in a standard cognitive control task to support motivation, usage time, usabil-ity, and therefore symptom reduction. In a previous pilot trial, we were able to document that de:)press® is superior to a non-gamified standard cognitive control training in reducing depression symptomatology. Based on these data, we now designed a full-size confirmatory trial for the pur-pose of testing the hypothesis that de:)press® provides a positive healthcare effect by means of reduction in depression severity compared to treatment as usual (TAU). In this randomized, con-trolled, clinical trial 112 patients will be randomized to the intervention group (IG) with de:)press® additional to TAU, or the control group (CG) receiving only TAU. For a period of 6 weeks, the IG is provided with de:)press®. To prove a stable efficacy of de:)press®, the primary endpoint is the dif-ference in the Montgomery-Åsberg Depression Scale (MADRS) change 4 weeks after the end of training between IG and CG.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, diverse,
* age >= 18,
* informed consent,
* sufficient understanding of German (native speaker or CEFR level B skills or higher),
* unipolar depression diagnosed according to ICD-10 (F32.0, F32.1, F32.2 or F33. 0, F32.1, F32.2).
* consultation with a physician due to depressive symptomatology within the last 6 months

Exclusion Criteria:

* Inability to give consent,
* inability to use de:)press® on a tablet or smartphone,
* acute suicidality,
* schizophrenia (F20),
* brief psychotic disorder (F23),
* schizoaffective disorder (F25),
* mental disorders due to known physiological conditions (F00 - F09),
* major depressive disorder, single episode, severe with psychotic features (F32.3),
* major depressive disorder, recurrent, severe with psychotic features (F33.3),
* Intellectual disability (F70 - F79).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
MADRS | 10 weeks
  Difference in symptom severity-reduction (MADRS) between IG and CG at the final examination.

SECONDARY OUTCOMES:
Response rate | 10 weeks
  Response rate (MADRS ≤ 50%) at the final examination.
Remission rate | 10 weeks
  MADRS score ≤ 10.
IDS-SR reduction | 10 weeks
  Reduction (IG vs. CG) of IDS-SR score during treatment phase and at final examination.
WHO-5 changes | 10 weeks
  Changes of well-being according to WHO-5 during treatment period and at final examination.
WPAI changes | 10 weeks
  Changes of functionality according to WPAI during treatment period and at final examination.
Training sessions | 6 weeks
  Number of completed training sessions in IG.
Adverse events | 10 weeks
  Adverse events.
Self-esteem | 10 weeks
  Influence of RSES on the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fallgatter, Prof., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided